CLINICAL TRIAL: NCT01328171
Title: An Open-label 2:1 Randomized Phase II Study of Panitumumab Plus FOLFOXIRI or FOLFOXIRI Alone as First-line Treatment of Patients With Non-resectable Metastatic Colorectal Cancer and RAS Wild Type
Brief Title: FOLFOXIRI With or Without Panitumumab in Metastatic Colorectal Cancer (VOLFI)
Acronym: VOLFI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Amgen (Industry); ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO KRK 0109; 2009-017731-17 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Folic Acid; Fluorouracil; Oxaliplatin; Irinotecan; FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (FOLFOXIRI + Panitumumab) (Experimental): FOLFOXIRI + Panitumumab
  Interventions: Drug: FOLFOXIRI + Panitumumab
- B (FOLFOXIRI) (Active Comparator): FOLFOXIRI
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI + Panitumumab — irinotecan 150 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 3000 mg/m² cont. inf. + panitumumab, iv, 6 mg/kg BW all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: Vectibix (Panitumumab); folic acid; 5-FU; oxaliplatin; irinotecan
  Arms: A (FOLFOXIRI + Panitumumab)
Drug: FOLFOXIRI — irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 3200 mg/m² cont. inf. all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: folic acid; 5-FU; oxaliplatin; irinotecan
  Arms: B (FOLFOXIRI)

SUMMARY:
The aim of the trial is to optimize response rates and rates of secondary resections of metastases in patients with initially non-resectable metastatic colorectal cancer of RAS wildtype. The patients will be treated in two therapy groups:

Experimental arm A: Chemotherapy with FOLFOXIRI + panitumumab Standard arm B: Chemotherapy with FOLFOXIRI

ELIGIBILITY:
Inclusion Criteria:

* Cohort I: Histologically confirmed and definitively inoperable or irresectable metastatic colorectal cancer. Focus on patients with large tumor load at metastatic sites and/or symptomatic metastatic disease
* Cohort II: Chance of secondary resection with curative intent defined and reviewed by expert panel
* Adult patients (≥ 18 years of age)
* RAS wild-type tested in

  * KRAS exon 2 (codons 12/13)
  * KRAS exon 3 (codons 59/61)
  * KRAS exon 4 (codons 117/146)
  * NRAS exon 2 (codons 12/13)
  * NRAS exon 3 (codons 59/61)
  * NRAS exon 4 (codons 117/146) assessed by an institution participating in and certified by the specific working group of the Deutsche Gesellschaft für Pathologie)
* At least one measurable lesion according to RECIST measured within 3 weeks prior to registration
* No previous chemotherapy for metastatic disease (adjuvant chemotherapy for non-metastatic disease is allowed if terminated more than 6 months ago)
* Performance status ECOG 0-1
* Male and female subjects > 18 years of age
* Adequate haematological, hepatic, renal and metabolic function parameters:

Leukocytes > 3000/mm³, ANC ≥ 1500/mm3, platelets ≥ 100,000/mm3, Hb > 9g/dl (may be transfused or treated with erythropoietin to maintain or exceed this level)Creatinine clearance ≥ 50 ml/min or serum creatinine ≤ 1.5 x upper limit of normal Bilirubin ≤ 1.5 x upper limit of normal, GOT-GPT ≤ 2.5 x upper limit of normal in absence of liver metastases, or ≤ 5 x upper limit of normal in presence of liver metastases, AP ≤ 5 x upper limit of normal Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal (may be substituted to maintain or exceed this level)

* Negative pregnancy test and willingness to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* Before subject registration, written informed consent must be given according to ICH-GCP, and national/local regulations.

Exclusion Criteria:

* Past or current history of malignancies except for the indication under this study and curatively treated:
* Basal and squamous cell carcinoma of the skin
* In-situ carcinoma of the cervix
* Other malignant disease without recurrence after at least 5 years of follow-up
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment.
* Clinically relevant interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* History of evidence upon physical examination of CNS disease unless adequately treated (e.g. primary brain tumour, seizure not controlled with standard medical therapy, brain metastases or history of stroke).
* Pre-existing neuropathy > grade 1 (NCI CTCAE), except for loss of tendon reflex
* Allogeneic transplantation requiring immunosuppressive therapy.
* Severe non-healing wounds, ulcers or bone fractions.
* Evidence of bleeding diathesis or coagulopathy.
* Patients not receiving therapeutic anticoagulation must have an INR < 1,5 ULN and aPTT < 1,5 ULN within 7 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of randomisation.
* Concomitant therapy with certain anti-viral medicines (sorivudine and brivudine or analogue compounds).
* Major surgical procedure, open biopsy, nor significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study except for surgery for colorectal cancer with curative intent and central venous line placement for chemotherapy administration.
* Pregnancy or breastfeeding women.
* Subjects with known allergy to the study drugs or to any of its excipients.
* Known DPD deficiency.
* Current or recent (within the 28 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
* Known grade III/IV allergic reaction against monoclonal antibodies.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
overall response rate | up to about 6 month
  RECIST

SECONDARY OUTCOMES:
overall response rate in each cohort | up to about 6 month
  RECIST
secondary resection rate with curative intent for patients cohort I | up to about 6 month
pathological response in liver surgery specimen | up to about 6 month
  metrics: Pathological complete response (pCR): no residual cancer cells;major response (pPR): 1% to 49% residual cancer cells remaining; minor response (pMR): 50% to 99% residual cancer cells remaining; no response (pNR): 100% residual cancer cells remaining
disease control rate | up to about 6 month
  CR + PR + SD rate according to RECIST
progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
duration of response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
  analyzed for responders only
time to response | up to about 6 month
overall survival | From date of randomization until the date of death from any cause assessed up to 4 years
time to recurrence (cohort II in case of secondary resection) | up to 4 years
toxicity and feasibility | up to about 6 month
  number of patients with adverse events and severity according to NCI CTC 3.0
liver toxicity for resected patients (central histological review); biopsies should be obtained for all patients pre-treatment | up to 1 year
  histological findings according to CASH/SOS scores
QL (QLQ C30) | Pre-treatment, before start of every 3rd cycle and at the end of treatment
  scores according to EORTC QLQ-C30 scoring manual (Quality of life)
translational research (EGFR genetics and proteomics): prognostic and predictive impact on efficacy outcomes | up to 4 years
  Determination of EGFR mutations (exons 18, 19, 20, 21) in tumor tissue; determination of PIK3CA mutations (exon 9, 20) in tumor tissue; determination of EGFR, ERCC1, TS, MTHFR, OPRT, DHFR and CDKN polymorphism from normal and tumor tissue; determination of ERCC1, PTEN and TS protein expression in tumor tissue; epigenetic candidates; further exploratory studies such as miRNA analysis as approved by the AIO review board

CONTACTS AND LOCATIONS:
Overall Officials: Michael Geißler, MD, PhD, Principal Investigator — Department of Oncology and Gastroenterology, Academic Teaching Hospital Esslingen
Locations (19):
- Germany (19):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - Ortenau Klinikum, Lahr, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Kreiskliniken Esslingen gGmbH Klinik Nürtingen, Nürtingen, Baden-Wurttemberg
  - Schwerpunktpraxis und Tagesklinik Onkologie Hämatologie Gastroenterologie Palliativmedizin Drs. Höring, Respondek, Schwinger, Thunert, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Ulm Zentrum für Innere Medizin, Ulm, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Leopoldina-Krankenhaus der Stadt Schweinfurth gGmbH, Schweinfurt, Bavaria
  - Klinikum der J.W. Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg, Hesse
  - Franziskus Hospital Niels-Stensen-Kliniken Klinik für Internistische Onkologie und Hämatologie, Georgsmarienhütte, Lower Saxony
  - Marienhospital Osnabrück Niels-Stensen-Kliniken Klinik für Innere Medizin, Osnabrück, Lower Saxony
  - St. Vincenz-Krankenhaus, Paderborn, North Rhine-Westphalia
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier, Rhineland-Palatinate
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Jena, Jena, Thuringia

REFERENCES:
- [Derived] Modest DP, Martens UM, Riera-Knorrenschild J, Greeve J, Florschutz A, Wessendorf S, Ettrich T, Kanzler S, Norenberg D, Ricke J, Seidensticker M, Held S, Buechner-Steudel P, Atzpodien J, Heinemann V, Seufferlein T, Tannapfel A, Reinacher-Schick AC, Geissler M. FOLFOXIRI Plus Panitumumab As First-Line Treatment of RAS Wild-Type Metastatic Colorectal Cancer: The Randomized, Open-Label, Phase II VOLFI Study (AIO KRK0109). J Clin Oncol. 2019 Dec 10;37(35):3401-3411. doi: 10.1200/JCO.19.01340. Epub 2019 Oct 14. PMID 31609637
- See also: AIO-Homepage — http://www.aio-portal.de